CLINICAL TRIAL: NCT04575610
Title: Investigation of IRAK4 Inhibition to Mitigate the Impact of COVID-19 in Severe SARS-CoV-2 (I-RAMIC)
Brief Title: IRAK4 Inhibition in Treatment of COVID-19 With ARDS (I-RAMIC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to lack of enrollment reflecting the decrease in number of COVID infections. There were no safety and/or efficacy concerns involved in the decision to stop enrollment.
Sponsor: Yale University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Hyung Chun, Associate Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2000028042
Record Dates: First submitted 2020-08-05; First posted 2020-10-05 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: COVID-19
Keywords: Protein Kinase Inhibitors; Enzyme Inhibitors; Molecular Mechanisms of Pharmacological Action
MeSH Terms: conditions — COVID-19 | interventions — 1-(((2S,3S,4S)-3-ethyl-4-fluoro-5-oxopyrrolidin-2-yl)methoxy)-7-methoxyisoquinoline-6-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PF-06650833 + Standard of Care (Experimental): Subjects randomized to the PF-06650833 arm of the study will receive 200 mg IR suspension formulation every 6 hours (via nasogastric [NG] tube, orogastric [OG] tube, or equivalent) if unable to take tablets by mouth (PO). All dosing of PF-06650833 will be in addition to current hospital SOC therapy.
  Interventions: Drug: PF-06650833
- Placebo + Standard of Care (Active Comparator): Matching placebo tablets will be administered.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-06650833 — Subjects randomized to the PF-06650833 arm of the study will receive 200 mg IR suspension formulation every 6 hours (via nasogastric [NG] tube, orogastric [OG] tube, or equivalent) if unable to take tablets by mouth (PO). Subjects for whom concomitant administration of a strong inhibitor of cytochrome P450 (CYP) 3A4 will have the dose of the IR formulation to 200 mg once daily (QD). Subjects who can take tablets PO will receive 400 mg PF-06650833 (2-200 mg tablets) of the MR formulation QD under fasted conditions (preferably at least 4 hours after and 1.5 hours before a meal). No dose adjustment is needed for subjects taking the MR tablet preparation, except if co-administered with ritonavir in which case the dose should be reduced to 200 mg MR QD. All dosing of PF-06650833 will be in addition to current hospital SOC therapy.
  Arms: PF-06650833 + Standard of Care
Drug: Placebo — Matching placebo tablets will be administered.
  Arms: Placebo + Standard of Care

SUMMARY:
The purpose of this study is to assess the efficacy of PF-06650833 in addition to standard-of-care compared to standard-of-care treatment alone in improving outcomes in patients with COVID-19.

DETAILED DESCRIPTION:
Proposed is a randomized, double-blind, placebo-controlled, parallel group Phase 2 study of the efficacy and safety of PF-06650833, an investigational drug, in hospitalized adult male and female patients with SARS-CoV-2-induced ARDS who need mechanical ventilation.

The primary objective of this study is to assess the efficacy of PF-06650833 in addition to standard-of-care compared to standard-of-care treatment alone in improving outcomes in patients with COVID-19, evidence of increased inflammation, and ARDS requiring mechanical ventilation or extracorporeal membrane oxygenation at time of admission.

The secondary objectives of this study are to evaluate:

1. Proportion of patients alive, extubated, and receiving no more that low flow oxygen supplementation by nasal cannula or face mask (excluding extubation for compassionate purposes in terminal patients). This would correspond to an at least 2-point improvement in the National Institute of Allergy and Infectious Diseases (NIAID) ordinal scale (1 = non hospitalized, no limitations on activity, and 8 = death) at Days 29 and 61
2. Proportion of patients alive, extubated, and receiving any level oxygen supplementation, including non-invasive positive pressure ventilation or high flow oxygen device (excluding extubation for compassionate purposes in terminal patients). This would correspond to an at least 1-point improvement in the NIAID ordinal scale (1 = non hospitalized, no limitations on activity, and 8 = death) at Days 29 and 61
3. Percentage of patients in each category of the NIAID 8-point ordinal scale of disease severity (Days 8, 15, 22, 29, and 61). The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows:

   * Not hospitalized, no limitations on activities;
   * Not hospitalized, limitation on activities and/or requiring home oxygen*
   * Hospitalized, not requiring supplemental oxygen* - no longer requires ongoing medical care
   * Hospitalized, not requiring supplemental oxygen* - requiring ongoing medical care (COVID-19 related or otherwise)
   * Hospitalized, requiring supplemental oxygen*;
   * Hospitalized, on non-invasive ventilation (NIV)** or high flow oxygen device;
   * Hospitalized, on invasive mechanical ventilation or ECMO;
   * Death

     * For patients on chronic home O2 supplementation, supplemental O2 is defined as >= home O2 requirement.

       * Use of NIV for chronic conditions [e.g. Obstructive sleep apnea (OSA)] is not applicable
4. Mortality rate at Day 61
5. Time to a 1-point improvement in the NIAID 8-point ordinal scale of disease severity
6. Time to a 2-point improvement in the NIAID 8-point ordinal scale of disease severity
7. Change from baseline in the ordinal scale from Day 1 to Days 3, 5, 8, 11, 15, 22, and
8. Arterial partial pressure of oxygen (PaO2) / Fractional concentration of inspired oxygen (FiO2) ratio (or P/F ratio)
9. Change of the Sequential Organ Failure Assessment (SOFA). The SOFA evaluates 6 variables, each representing an organ system (one for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems), and scored from 0 (normal) to 4 (high degree of dysfunction/failure). Thus, the maximum score may range from 0 to 24.
10. Duration (days) of mechanical ventilation
11. Ventilator free days
12. Safety as assessed by reporting of adverse events (AEs), changes in clinical laboratory parameters (e.g., haemoglobin (Hb), white blood cell (WBC) count, platelets, hepatic transaminases, bilirubin, serum creatinine)

ELIGIBILITY:
INCLUSION CRITERIA

1. Adult male and female patients, including women of childbearing potential, at least 18 years of age, inclusive
2. Participant (or legally authorized representative) capable of giving signed informed consent
3. Laboratory-confirmed novel coronavirus (SARS-CoV-2) infection
4. Clinical findings and an imaging study consistent with ARDS;
5. PaO2 / FiO2 ratio < 300;
6. A requirement for mechanical ventilation ≤ 48 hours prior to enrollment.
7. Evidence of increased inflammation as assessed by hsCRP > ULN AND at least ONE of the following being > upper limit of normal (as available):

   1. ferritin
   2. procalcitonin
   3. D-dimer
   4. fibrinogen
   5. LDH
   6. PT/PTT

EXCLUSION CRITERIA

1. Suspected or known active systemic bacterial, viral (except SARS-CoV2 infection), or fungal infections
2. Active herpes zoster infection
3. Known active or latent tuberculosis (TB) or history of inadequately treated TB
4. Active hepatitis B or hepatitis C
5. Known history of human immunodeficiency virus (HIV) infection with a detectable viral load or CD4 count < 500 cells / mm3 (patients for whom documented viral load or CD4 counts are available will be excluded)
6. Active hematologic cancer
7. Metastatic or intractable cancer
8. Pre-existing neurodegenerative disease
9. Severe hepatic impairment defined as Child-Pugh Class B or Class C at baseline
10. Severe renal impairment with an estimated glomerular filtration rate (eGFR) < 45 mL/min/1.73 m2
11. Severe anemia (Hb < 8.0 g/dL)
12. Any of the following abnormal laboratory values:

    1. absolute lymphocyte count <250 cells/mm3
    2. absolute neutrophil Count (ANC) <1000 cells/mm3
    3. Platelet count <50,000 cells/mm3
    4. ALT or AST > 5X ULN, or other evidence of hepatocellular synthetic dysfunction or total bilirubin > 2X ULN
13. Any other medical condition or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study
14. Prohibited concomitant therapy (see section 1.12.7.2)
15. Pregnancy (a negative urine or serum pregnancy test is required for inclusion)
16. Immunocompromised patients, patients with known immunodeficiencies or taking potent immunosuppressive agents (e.g., azathioprine, cyclosporine)
17. Anticipated survival < 72 hours as assessed by the Investigator.
18. Participation in other clinical trials of investigational treatments for COVID-19
19. Known history of nephrolithiasis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-11-27 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2021-10-06 (Actual)

PRIMARY OUTCOMES:
All-cause mortality at Day 29 | Up to 29 days
  All-cause mortality at Day 29 (end of planned treatment period).

SECONDARY OUTCOMES:
Disease Severity (8 point scale) | 29 days
  Proportion of patients alive, extubated, and receiving no more than low flow oxygen supplementation by nasal cannula or face mask (excluding extubation for compassionate purposes in terminal patients). This would correspond to an at least 2 point decrease in the NIAID ordinal scale. The NIAID scale is as follows:
  1. Not hospitalized, no limitations on activities
  2. Not hospitalized, limitations on activities and/or requiring home oxygen
  3. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care
  4. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise)
  5. Hospitalized, requiring supplemental oxygen
  6. Hospitalized, on non-invasive ventilation or high-flow oxygen devices
  7. Hospitalized, on invasive mechanical ventilation or ECMO
  8. Death
Disease Severity (8 point scale) | 61 days
  Proportion of patients alive, extubated, and receiving no more than low flow oxygen supplementation by nasal cannula or face mask (excluding extubation for compassionate purposes in terminal patients). This would correspond to an at least 2 point decrease in the NIAID ordinal scale (1 = not hospitalized, no limitations on activities, and 8 = death) at Day 61.
Disease Severity (8 point scale) | 29 days
  Proportion of patients alive, extubated, and receiving any level oxygen supplementation, including non-invasive positive pressure ventilation or high flow oxygen device (excluding extubation for compassionate purposes in terminal patients). This would correspond to an at least 1-point decrease in the NIAID ordinal scale (1 = not hospitalized, no limitations on activities, and 8 = death) at Day 29.
Disease Severity (8 point scale) | 61 days
  Proportion of patients alive, extubated, and receiving any level oxygen supplementation, including non-invasive positive pressure ventilation or high flow oxygen device (excluding extubation for compassionate purposes in terminal patients). This would correspond to an at least 1-point decrease in the NIAID ordinal scale (1 = not hospitalized, no limitations on activities, and 8 = death) at Day 61.
Disease Severity (8 point scale) | 8 days
  Percentage of patients in each category of the NIAID 8-point ordinal scale of disease severity at Day 8. The ordinal scale is an assessment of the clinical status at the first assessment of a given study day in which 1 = not hospitalized, no limitations on activities, and 8 = death.
Disease Severity (8 point scale) | 15 days
  Percentage of patients in each category of the NIAID 8-point ordinal scale of disease severity at Day 15. The ordinal scale is an assessment of the clinical status at the first assessment of a given study day in which 1 = not hospitalized, no limitations on activities, and 8 = death.
Disease Severity (8 point scale) | 22 days
  Percentage of patients in each category of the NIAID 8-point ordinal scale of disease severity at Day 22. The ordinal scale is an assessment of the clinical status at the first assessment of a given study day in which 1 = not hospitalized, no limitations on activities, and 8 = death.
Disease Severity (8 point scale) | 29 days
  Percentage of patients in each category of the NIAID 8-point ordinal scale of disease severity at Day 29. The ordinal scale is an assessment of the clinical status at the first assessment of a given study day in which 1 = not hospitalized, no limitations on activities, and 8 = death.
Disease Severity (8 point scale) | 61 days
  Percentage of patients in each category of the NIAID 8-point ordinal scale of disease severity at Day 61. The ordinal scale is an assessment of the clinical status at the first assessment of a given study day in which 1 = not hospitalized, no limitations on activities, and 8 = death.
Mortality | 61 days
  Mortality rate at day 61
Disease Severity (8 point scale) | 29 days
  Time to a 1-point decrease in the NIAID 8-point ordinal scale of disease severity (1 = not hospitalized, no limitations on activities, and 8 = death).
Disease Severity (8 point scale) | 29 days
  Time to a 2-point decrease in the NIAID 8-point ordinal scale of disease severity.
Disease Severity (8 point scale) | 3 days
  Change from baseline in the ordinal scale from Day 1 to Days 3.
Disease Severity (8 point scale) | 5 days
  Change from baseline in the ordinal scale from Day 1 to Days 5.
Disease Severity (8 point scale) | 8 days
  Change from baseline in the ordinal scale from Day 1 to Days 8.
Disease Severity (8 point scale) | 11 days
  Change from baseline in the ordinal scale from Day 1 to Days 11.
Disease Severity (8 point scale) | 15 days
  Change from baseline in the ordinal scale from Day 1 to Days 15.
Disease Severity (8 point scale) | 22 days
  Change from baseline in the ordinal scale from Day 1 to Days 22.
Disease Severity (8 point scale) | 29 days
  Change from baseline in the ordinal scale from Day 1 to Days 29.
P/F ratio | Up to 29 days
  PaO2 (partial pressure of oxygen) / FiO2 (fraction of inspired oxygen, FiO2) ratio (or P/F ratio)
Change of the SOFA score. | Up to 29 days
  The SOFA evaluates 6 variables, each representing an organ system (one for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems), and scored from 0 (normal) to 4 (high degree of dysfunction/failure). Thus, the maximum score may range from 0 to 24.
Duration (days) of mechanical ventilation | Up to 29 days
  The duration is days spent on mechanical ventilation.
Ventilator free days. | Up to 29 days
  The number of days hospitalized not on a ventilator.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Up to 29 days

CONTACTS AND LOCATIONS:
Overall Officials: Hyung Chun, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No